CLINICAL TRIAL: NCT03687190
Title: Integrative Medicine and Tai-chi in Clinical Status of Spinocerebellar Ataxia
Brief Title: Could Tai-chi Help Maintain Balance of Spinocerebellar Ataxia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Chiu Chung Min, Adjunct Physician, Changhua Christian Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 121013
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Spinocerebellar Ataxias; Tai Chi
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai chi (Experimental): participants in this group accepted Tai chi exercise and conventional medicine.
  Interventions: Behavioral: Tai chi; Drug: conventional medicine
- controlled group (Active Comparator): participants were not received Tai chi exercise, but only routine conventional medicine
  Interventions: Drug: conventional medicine

INTERVENTIONS:
Behavioral: Tai chi — participants were required to receive hospital-based Tai chi training at least once a month, and home-based Tai chi exercise at least three times a week over the next 9 months
  Arms: Tai chi
Drug: conventional medicine — participants without Tai chi training still received routine conventional medicine

SUMMARY:
Spinocerebellar atrophy is the most common autosomal dominant inherited ataxia. There are over thirty subtypes, which characterize neurologic features differently. They all have obvious substantial cerebellar atrophies in image, and unstable gait、ataxia. In general a prevalence of about three cases per 100 000 people is assumed, but this may be an underestimate. Progressive neurologic degeneration, in about 10-20 years, will leads to disability or wheelchair-dependent. Accompanying with fatigue, downhill course of the disease often made patients depressive and hopeless. The recent review of researches concludes no effective therapy for the disease. The purpose of the investigator's study is to explore the Tai-chi exercise effect for spinocerebellar ataxia.

ELIGIBILITY:
Inclusion Criteria:

* progressive ataxia accompanied with the observation of cerebellar atrophy on magnetic resonance or computed tomography images
* SARA score of less than 20

Exclusion Criteria:

* Patients with complicated cerebellar disorders, such as multiple system atrophy, Parkinson-plus syndromes, secondary cerebellar degeneration from encephalitis, trauma, hypoxia, cerebrovascular diseases, and toxic- or drug-induced cerebellar degeneration
* SARA score of larger than 20

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Chien Lo, Principal Investigator — Director of Chinese Medicine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tai Chi: participants in this group accepted Tai chi exercise and conventional medicine.
  Tai chi: participants were required to receive hospital-based Tai chi training at least once a month, and home-based Tai chi exercise at least three times a week over the next 9 months conventional medicine: participants without Tai chi training still received routine conventional medicine
- Controlled Group: participants were not received Tai chi exercise, but only routine conventional medicine conventional medicine: participants without Tai chi training still received routine conventional medicine
Period: Overall Study
Arm/Group | Tai Chi | Controlled Group
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tai Chi: Subjects accepted Tai Chi exercise once a week in the hospital, and home-based training with a video.
- Controlled Group: No Tai Chi training. Only regular out-patient clinic visiting.
- Total: Total of all reporting groups
Arm/Group | Tai Chi | Controlled Group | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51.5 [43.75 to 60] | 51 [32 to 55] | 51 [40 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 6 | 6 | 12
scale for assessment and rating of ataxia [Median (Inter-Quartile Range); unit: units on a scale] — Scale for assessment and rating of ataxia (SARA) is used to assess patients of ataxia worldwide. It contains eight aspects, including gait, standing, sitting, finger-nose-finger test, heel to shin, and etc.. It is also an appropriate measure tool for longitudinal assessment of disease progression. The score ranges from 0 to 40 points, while higher points means worse ataxia.
  units on a scale | 9 [7.75 to 10] | 9.5 [6 to 13] | 9.5 [7 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Scale for the Assessment and Rating of Ataxia(SARA)
Description: SARA assesses eight aspects of cerebellar function: walking, sitting, standing, speaking, finger chasing, the nose-finger test, fast alternating hand movements, and the heel-shin slide. The eight categories accumulate score ranging from 0 (no ataxia) to 40 (most severe ataxia).Gait (0-8 points),Stance (0-6 points),Sitting (0-4 points),Speech disturbance (0-6 points),Finger chase (0-4 points),Nose-finger test (0-4 points),Fast alternating hand movement (0-4 points),Heel-shin slide (0-4 points)
Time Frame: assessed at baseline and 9 months, 9 months reported as Outcome Measure Data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Tai Chi: Subjects accepted Tai Chi exercise once a week in the hospital, and home-based training with a video. We measured the SARA before and after the nine months.
- Controlled Group: No Tai Chi training. Only regular out-patient clinic visiting. We measured the SARA before and after the nine months.
Arm/Group | Tai Chi | Controlled Group
Number analyzed (Participants) | 12 | 9
score on a scale | 11.5 [8.5 to 12.5] | 9 [7 to 12.5]

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Controlled Group: Participants without Tai chi training still received routine conventional medicine
Arm/Group | Tai Chi | Controlled Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

LIMITATIONS AND CAVEATS:
There were insufficient case numbers in this study, in both groups. There were patients with different gene types, non-hereditary, or even multiple system atrophy in the recruited subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No